CLINICAL TRIAL: NCT01128049
Title: Non-invasive Tear Film Dynamic Measurements in Normal, MGD (Meibomium Gland Dysfunction) and Aqueous Deficient Dry Eye(ADDE) Subjects After Saline Instillation
Brief Title: Non-invasive Tear Film Dynamic Measurements in Normal, MGD and ADDE Subjects After Saline Instillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, James V. Aquavella, MD, Medical Doctor and Department Faculty, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B&L 32280
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Aqueous Deficient Dry Eye; Meibomium Gland Dysfunction
Keywords: Aqueous deficient dry eye (ADDE); Meibomium Gland Dysfunction (MGD); Normal/Control (Non Dry Eye)
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal Patient Population (Active Comparator): Non-Dry Eye patient population (intervention remains the same across all arms)
  Interventions: Behavioral: Subjective Questionnaire; Procedure: Measurement with wavefront sensor (right eye, then left eye); Drug: Instill Saline Drop
- MGD Patient Population (Active Comparator): Meibomium Gland Dysfunction population(intervention remains the same across all arms)
  Interventions: Behavioral: Subjective Questionnaire; Procedure: Measurement with wavefront sensor (right eye, then left eye); Drug: Instill Saline Drop
- ADDE Population (Active Comparator): Aqueous Deficient Dry Eye population(intervention remains the same across all arms)
  Interventions: Behavioral: Subjective Questionnaire; Procedure: Measurement with wavefront sensor (right eye, then left eye); Drug: Instill Saline Drop

INTERVENTIONS:
Behavioral: Subjective Questionnaire — The team will use a one page questionnaire to obtain subjective input before the first set of measurements and after instilling the Saline drop.
Procedure: Measurement with wavefront sensor (right eye, then left eye) — The wavefront instrument measures the eye's ability to create a sharp image by briefly shining a laser light from the wavefront sensor into the eye and measuring the light that bounces back through the cornea. For these measurements, subjects will sit on a chair and be instructed to place their chin in a chin rest and lean their forehead against a forehead rest. The subject will be instructed to hold his/her head steady, look in a certain direction, blink or not blink. We will obtain the measurements over a short period of up to approximately 45 seconds. We will start recording data asking the subject to either blink naturally or to hold his/her eye open for a few (up to 10) seconds, and repeat the blink and hold sequence usually for up to four times.
Drug: Instill Saline Drop — One drop will be instilled in both eyes and patient will wait 5 minutes prior to repeating the questionnaire and wavefront sensor. A single drop is approximately 30 µL and will be placed into the inferior cul-de-sac while the patient looks up.
  Other Names: Ocufresh eye wash

SUMMARY:
Compare the objective tear film dynamic measurements in three different populations (MGD [Meibomium Gland Dysfunction], ADDE [Aqueous Deficient Dry Eye] and normal/control [non-dry eye]) and the subjective experience before and after instilling a single drop of saline in each eye.

Currently available office-based tests for dry eye do not reliably correlate with patients' subjective symptoms. This study is interested in assessing how individuals with these two different ocular surface diseases compare with the normal population when measured objectively using two different instruments.

DETAILED DESCRIPTION:
There will be one study day with a single visit that will consist of taking two sets of measurements. Baseline measurements are taken in both eyes using a wavefront sensor to measure visual quality followed by saline instillation. Five minutes after drops, visual quality is again measured to evaluate changes in tear dynamics.

ELIGIBILITY:
General Inclusion Criteria:

* Good general Health
* The subject must appear able and willing to adhere to the instructions set forth in this protocol (such as not use warm compresses or artificial tears/lubricant or excessive eye makeup before the visit on the study day).

General Exclusion Criteria:

* Ocular disease, infection or inflammation (allergy, blepharitis) that is clinically significant (grade 3 or 4) that in the opinion of the PI would not be a good subject.
* Systemic disease or use of medication that in the opinion of the PI would not be a good subject.
* Infectious diseases (e.g. hepatitis, tuberculosis) or an immuno-suppressive disease (e.g. HIV).
* Contact lens wearer.
* Pregnancy or lactation.
* Diabetes.
* Inclusion or exclusion criteria of the other cohorts.

Cohort Specific Inclusion Criteria:

* ADDE cohort: Schirmer I < 10 mm, BUT ¬< 5 seconds, Fluorescein 0 or 1, currently using an artificial tear for ocular comfort at least occasionally.
* MGD cohort: Diagnosis of moderate or severe MGD
* Normal/Control (Non Dry-Eye): meets general inclusion and exclusion criteria

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James V Aquavella, MD, Principal Investigator — University of Rochester
Locations (1):
- The Flaum Eye Institute-University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Patient Population: Subjects with no symptoms and no diagnosis of dry eye. Schirmer's value ≥ 10mm/5 mins and a fluorescein tear break-up time >5 secs with no surface staining.
- MGD Patient Population: Subjects with a meibomian gland dysfunction on a slitlamp examination with a fluorescein tear break-up time <5 secs.
- ADDE Population: Subjects with schirmer's value < 10mm/5 mins and no meibomian gland dysfunction.
Period: Overall Study
Arm/Group | Normal Patient Population | MGD Patient Population | ADDE Population
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Patient Population | MGD Patient Population | ADDE Population | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 15
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5 | 10
  Male | 2 | 3 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Visual Quality
Description: Average visual quality change over a 5 second blink cycle caused by movement of the tears over the surface of the eye by measuring optical irregularities.
Time Frame: 5 seconds
Population: The comparison was between normal, non-dry eye participants and dry eye groups.
Measure: Mean (Standard Deviation); unit: microns
Groups:
- Normal: Normal group included non-dry eye subjects.
- Meibomian Gland Dysfunction (MGD): Subjects with mild to moderate Meibomian Gland Dysfunction (MGD) on a slit lamp examination were included in this group.
- Aqueous Deficiency Dry Eye (ADDE): Subjects with a low tear volume measured by Schimer's score of less than 10 mm were included in this group.
Arm/Group | Normal | Meibomian Gland Dysfunction (MGD) | Aqueous Deficiency Dry Eye (ADDE)
Number analyzed (Participants) | 5 | 5 | 5
microns
  Visual Quality at Baseline | 0.3 (0.07) | 0.32 (0.08) | 0.19 (0.06)
  Visual Quality at 5 minutes after Saline | 0.3 (0.08) | 0.33 (0.08) | 0.23 (0.05)

ADVERSE EVENTS:
Time Frame: Over 1 year
Description: No Adverse Events were reported.
Arm/Group | Normal Patient Population | MGD Patient Population | ADDE Population
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor review required before publishing results.